CLINICAL TRIAL: NCT01475526
Title: El Valor de Nuestra Salud (The Value of Our Health)
Brief Title: The Value of Our Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guadalupe X. Ayala, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA140326 (NIH); 5R01CA140326-02 (NIH)
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Prevention of Chronic Disease; Prevention and Control; Diet
Keywords: grocery store; nutrition; Latino; Hispanic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): El Valor de Nuestra Salud Store Intervention
  Interventions: Other: El Valor de Nuestra Salud Store Intervention
- Control (No Intervention): No intervention. Business as usual

INTERVENTIONS:
Other: El Valor de Nuestra Salud Store Intervention — Changes to physical and social environment of grocery stores through implementation of the El Valor de Nuestra Salud intervention.
  Arms: Intervention

SUMMARY:
El Valor de Nuestra Salud [The Value of Our Health] is a 5-year study (2010-2014) involving grocery stores in San Diego County funded by the National Cancer Institute. The purpose of the study is to determine whether an in-store program can promote healthy foods through grocery stores. Sixteen stores in San Diego County will participate in El Valor de Nuestra Salud. The stores that participate in this study will be randomly assigned to either the intervention (program and evaluation) or control (evaluation only) group. We will test various strategies to promote healthy food shopping among customers of small-to-medium size Latino/Hispanic grocery stores. These strategies include changes to the store environment, food marketing efforts, and training of sales associates. Our evaluation protocol will determine whether the project is successful at improving aspects of the store and the employees, as well as whether customers shop for and eat healthier food products. The primary aim of the study is to evaluate the impact of the El Valor de Nuestra Salud intervention on consumption of fruits and vegetables among store customers.

DETAILED DESCRIPTION:
El Valor de Nuestra Salud [The Value of Our Health] is a 5-year study (2010-2014) involving grocery stores in San Diego County funded by the National Cancer Institute. The purpose of the study is to determine whether an in-store program can promote healthy foods through grocery stores. Sixteen stores in San Diego County participated in El Valor de Nuestra Salud. The stores that participated in this study were randomly assigned to either the intervention (program and evaluation) or control (evaluation only) group. We tested various strategies to promote healthy food shopping among customers of small-to-medium size Latino/Hispanic grocery stores. These strategies included changes to the store environment, food marketing efforts, and training of sales associates. Our evaluation protocol is designed to determine whether the project was successful at improving aspects of the store and the employees, as well as whether customers shop for and eat healthier food products. Customers were recruited as they enter the store to participate in project interviews and objective weight measures at baseline, 6-months post-baseline, and 12-months post-baseline. The primary aim of the study is to evaluate the impact of the El Valor de Nuestra Salud intervention on consumption of fruits and vegetables among store customers.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must be one of the main food shoppers of the household
* Must shop at study store at least once per week
* Must already be a purchaser of food products from this store
* Must be Latino
* Must speak Spanish and/or English
* Must be able to read in Spanish
* Must eat 4 or less cups of fruits and vegetables per day
* Must plan on living in San Diego County for at least the next 12 months

Exclusion Criteria:

* Must not have any dietary restrictions limiting consumption of fruits and vegetables
* Participating customers cannot shop at other study stores in that wave more than once a month
* Participating customers cannot shop at intervention stores from previous waves more than once a month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in fruit and vegetable consumption of store customers from baseline to 6-months as assessed by the NCI fruit and vegetable screener | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe X Ayala, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University Research Foundation, San Diego, California, United States

REFERENCES:
- [Derived] Stuber JM, Beulens JW, Ayala GX, Crozier SR, Dijkstra SC, Lin SF, Vogel C, Mackenbach JD. Can nudge interventions targeting healthy food purchases in real-world grocery stores reduce diet-related health disparities? A pooled analysis of four controlled trials. Int J Behav Nutr Phys Act. 2024 Dec 3;21(1):137. doi: 10.1186/s12966-024-01687-3. PMID 39627771
- [Derived] Ayala GX, Pickrel JL, Baquero B, Sanchez-Flack J, Lin SF, Belch G, Rock CL, Linnan L, Gittelsohn J, Ji M, Elder JP, Mayer J. The El Valor de Nuestra Salud clustered randomized controlled trial store-based intervention to promote fruit and vegetable purchasing and consumption. Int J Behav Nutr Phys Act. 2022 Feb 17;19(1):19. doi: 10.1186/s12966-021-01220-w. PMID 35177070
- See also: El Valor de Nuestra Salud is housed within the Institute for Behavioral and Community Health at SDSU — http://www.ibachsd.org/